CLINICAL TRIAL: NCT00031694
Title: A Phase II Study of Sequential Paclitaxel and Bryostatin-1 for Patients With Advanced Pancreatic Cancer
Brief Title: Paclitaxel and Bryostatin 1 in Treating Patients With Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03003; 01-09-224 (Other: Montefiore Medical Center); NCI-5624 (Other: CTEP); N01CM17103 (NIH)
Record Dates: First submitted 2002-03-08; First posted 2003-01-27 (Estimated); Results first posted 2015-04-21 (Estimated); Last update posted 2021-06-11 (Actual); Status verified 2021-05

CONDITIONS: Acinar Cell Adenocarcinoma of the Pancreas; Duct Cell Adenocarcinoma of the Pancreas; Recurrent Pancreatic Cancer; Stage III Pancreatic Cancer; Stage IV Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Paclitaxel; Taxes; bryostatin 1; Bryostatins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (paclitaxel, bryostatin 1) (Experimental): Patients receive paclitaxel IV over 1 hour on day 1 followed by bryostatin 1 IV over 1 hour on day 2 of weeks 1-3. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: paclitaxel; Drug: bryostatin 1

INTERVENTIONS:
Drug: paclitaxel — Given IV
  Other Names: Anzatax; Asotax; TAX; Taxol
Drug: bryostatin 1 — Given IV
  Other Names: B705008K112; BRYO; Bryostatin

SUMMARY:
Phase II trial to study the effectiveness of combining paclitaxel and bryostatin-1 in treating patients who have locally advanced unresectable or metastatic pancreatic cancer. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Bryostatin-1 may help paclitaxel kill more cancer cells by making tumor cells more sensitive to the drug.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the response rates to weekly, sequential paclitaxel/ bryostatin-1 in patients with unresectable and metastatic pancreatic cancer.

II. To determine the toxicity of therapy. III. To determine patient survival after therapy. IV. To determine Bryostatin-1 pharmacokinetics.

OUTLINE: This is an open-label, multicenter study.

Patients receive paclitaxel IV over 1 hour on day 1 followed by bryostatin 1 IV over 1 hour on day 2 of weeks 1-3. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Histologic proof of adenocarcinoma of the pancreas that is locally advanced and considered surgically not resectable or metastatic
* Patients with or without prior treatment are eligible for treatment on protocol; prior treatment may have included one treatment course of chemo/RT and/ or one course of chemotherapy, but not two prior courses of chemotherapy;
* Measurable disease
* ECOG performance status of 0-1
* Ability to sign an informed consent form indicating awareness of the investigational nature of this study, in keeping with the policies of the hospital
* Patients may not be receiving any other concurrent chemotherapy, immunotherapy, or radiotherapy; the most recent treatment for pancreatic cancer, within the limitations of allowed prior therapy must be 28 days or longer prior to enrollment on study
* Absolute granulocytes > 1,500/mm^3
* Platelets > 150,000/mm^3
* Serum bilirubin < 1.5 mg/dl
* Serum creatinine < 1.5 mg/dl

Exclusion Criteria:

* Presence of any ongoing toxic effect from prior treatment
* Brain metastases
* History of active angina or myocardial infarction within 6 months; history of significant ventricular arrhythmia requiring medication with antiarrhythmics; well controlled atrial fibrillation on standard management will be permitted
* Pregnant or lactating women
* Pre-existing neurotoxicity that is graded 3+ or greater
* Serious intercurrent infections, or nonmalignant medical illnesses that are uncontrolled or whose control may be jeopardized by the complications of this therapy
* Psychiatric disorders rendering patients incapable of complying with the requirements of the protocol
* HIV infection
* Any other medical condition or reason that, in the investigator's opinion, makes the patient unsuitable to participate in a clinical trial (for example a history of prior poor compliance with treatment)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2002-03; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Kaubisch, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

REFERENCES:
- [Result] Lam AP, Sparano JA, Vinciguerra V, Ocean AJ, Christos P, Hochster H, Camacho F, Goel S, Mani S, Kaubisch A. Phase II study of paclitaxel plus the protein kinase C inhibitor bryostatin-1 in advanced pancreatic carcinoma. Am J Clin Oncol. 2010 Apr;33(2):121-4. doi: 10.1097/COC.0b013e3181a31920. PMID 19738452

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 19 patients were enrolled from 5 centers between March 2002 and October 2003.
Groups:
- Treatment (Paclitaxel, Bryostatin 1): Patients receive paclitaxel IV over 1 hour on day 1 followed by bryostatin 1 IV over 1 hour on day 2 of weeks 1-3. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
  paclitaxel: Given IV
  bryostatin 1: Given IV
  pharmacological study: Correlative studies
Period: Overall Study
Arm/Group | Treatment (Paclitaxel, Bryostatin 1)
Started | 19
Completed | 0
Not Completed | 19
Not completed — Adverse Event | 12
Not completed — Death | 2
Not completed — Withdrawal by Subject | 5

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Paclitaxel, Bryostatin 1)
Number analyzed (Participants) | 19
Age, Continuous [Median (Full Range); unit: years] | 56.0 [21 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 12
Race/Ethnicity, Customized [Number; unit: participants]
  Non-Hispanic whites | 13
  Non-Hispanic black | 3
  Hispanic | 3

OUTCOME MEASURES:

1. Primary Outcome: Response Rate of at Least 30%
Description: Number of participants with a Response rate of at least 30%. Response was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST).
Time Frame: Up to 8 years
Population: data not met
Measure: Number; unit: participants
Arm/Group | Treatment (Paclitaxel, Bryostatin 1)
Number analyzed (Participants) | 19
participants | 0

2. Secondary Outcome: Number of Participants With Adverse Events
Time Frame: Up to 8 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Paclitaxel, Bryostatin 1)
Number analyzed (Participants) | 19
Participants | 10

3. Secondary Outcome: Overall Survival
Description: Computed using the Kaplan-Meier estimator.
Time Frame: Up to 8 years
Population: Patients with locally advanced or metastatic pancreatic adenocarcinoma received a total of 52 cycles of therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Paclitaxel, Bryostatin 1)
Number analyzed (Participants) | 19
Participants | 17

4. Other Pre Specified Outcome: Bryostatin 1 Pharmacokinetics
Description: Not done-study terminated early
Time Frame: Week 1
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Treatment (Paclitaxel, Bryostatin 1)
Serious Adverse Events (participants affected / at risk) | 10/19
Other Adverse Events (participants affected / at risk) | 7/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Paclitaxel, Bryostatin 1) (N=19)
Leukopenia (Blood and lymphatic system disorders) | 5
Anemia (Blood and lymphatic system disorders) | 2
Death (General disorders) | 2
Abdominal pain (General disorders) | 2
Infection (Infections and infestations) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Thrombosis/embolism (Vascular disorders) | 2
Hemorrhage (Vascular disorders) | 2
ALT/SGPT (Hepatobiliary disorders) | 2
AST/SGOT (Hepatobiliary disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Paclitaxel, Bryostatin 1) (N=19)
Leukopenia (Blood and lymphatic system disorders) | 1
Anemia (Blood and lymphatic system disorders) | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 7
Abdominal pain (General disorders) | 3
Infection (Infections and infestations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less